CLINICAL TRIAL: NCT01874340
Title: A Phase II, Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Adaptive Dose-ranging Study to Evaluate the Efficacy and Safety of AIN457 (Secukinumab) in Patients With Relapsing Multiple Sclerosis
Brief Title: Efficacy and Safety of AIN457 (Secukinumab) in Patients With Relapsing Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early based upon development of another anti-IL17 fully human monoclonal antibody with better potential for treating MS patients
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457B2203; 2012-004019-29 (EudraCT Number)
Record Dates: First submitted 2013-05-28; First posted 2013-06-11 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Multiple Sclerosis; AIN457; Secukinumab; Magnetic Resonance Imaging; Relapsing Remitting Multiple Sclerosis; Autoimmune Diseases; Nervous System Diseases; Immune System Diseases; Demyelinating Diseases
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Autoimmune Diseases; Nervous System Diseases; Immune System Diseases; Demyelinating Diseases | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AIN457 low dose (Experimental): AIN457 will be administered intravenously. Approximately 65 patients will be randomized to AIN457 low dose in Stage 1. An additional 40 patients may be randomized to this group if it is one of the two selected dose groups to be expanded for Stage 2 following an Interim Analysis.
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator): Matching placebo will be administered intravenously. Approximately 105 patients will be randomized to placebo (65 in Stage 1 and 40 in Stage 2).
  Interventions: Drug: Placebo
- AIN457 middle dose (Experimental): AIN457 will be administered intravenously. Approximately 65 patients will be randomized to AIN457 middle dose in Stage 1. An additional 40 patients may be randomized to this group if it is one of the two selected dose groups to be expanded for Stage 2 following an Interim Analysis
  Interventions: Drug: AIN457
- AIN457 high dose (Experimental): AIN457 will be administered intravenously. Approximately 65 patients will be randomized to AIN457 high dose in Stage 1. An additional 40 patients may be randomized to this group if it is one of the two selected dose groups to be expanded for Stage 2 following an Interim Analysis.
  Interventions: Drug: AIN457

INTERVENTIONS:
Drug: Placebo — Placebo will be administered at predefined visits over the 6-month treatment phase.
  Arms: Placebo
Drug: AIN457 — AIN457 will be administered at predefined visits over the 6-month treatment phase.
  Arms: AIN457 high dose; AIN457 low dose; AIN457 middle dose

SUMMARY:
To evaluate the efficacy and safety of AIN457 versus placebo in patients with relapsing multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis according to 2010 revised McDonald criteria
* Disease duration of 10 years or less
* At least one relapse in the last year
* EDSS score 0 to 5.0 at entry

Exclusion Criteria:

* Active chronic disease of the immune system other than multiple sclerosis
* History of malignancy within the past 5 years
* Active systemic bacterial, viral or fungal infections
* Previous treatment with more than one class of multiple sclerosis therapies except for previous treatment with glatiramer acetate and interferon-beta(s)
* Any medically unstable condition
* Unable to undergo MRI scans or repeated blood tests
* Pregnant or nursing females
* Women of child-bearing potential must use reliable forms of contraception
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Novartis Investigative Site, Bruges, Belgium
- Novartis Investigative Site, Jihlava, Czechia
- Novartis Investigative Site, Saint-Herblain, France
- Novartis Investigative Site, Roma, RM, Italy
- Novartis Investigative Site, Osaka, Osaka, Japan
- Poland (2):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (2):
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Atakum / Samsun, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 15 mg/kg; AIN457 7 mg/kg; AIN457 3 mg/kg: AIN457 will be administered intravenously at day1, Week 2, week 4 and every 4 weeks therafter.
- Placebo: Matching placebo will be administered intravenously at day1, Week 2, week 4 and every 4 weeks therafter.
Period: Overall Study
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Started | 6 | 8 | 8 | 6
Completed | 0 | 0 | 0 | 1
Not Completed | 6 | 8 | 8 | 5
Not completed — Study terminated by Sponsor | 6 | 8 | 8 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.8 (7.73) | 34.5 (8.64) | 35.5 (9.71) | 34.0 (9.30) | 33.5 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 6 | 4 | 18
  Male | 2 | 4 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of New Gadolinium [Gd]-Enhancing T1-weighted Lesions
Description: Due to early termination this trial was not powered for efficacy no statistical analysis was performed
Time Frame: Months 3, 4, 5, 6
Population: Due to the early termination of the study and just one patient completing treatment as planned, no statistical analyses could be performed for the efficacy endpoints defined in the protocol.
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Annualized Relapse Rate
Description: Due to early termination this trial was not powered for efficacy no statistical analysis was performed
Time Frame: 6 Months
Population: as for outcome 1
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Combined Unique Active Lesions (CUAL)
Description: Due to early termination this trial was not powered for efficacy no statistical analysis was performed
Time Frame: Months 3, 4, 5, 6
Population: as for outcome 1
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Total Volume of T2-weighted Lesions
Description: Due to early termination this trial was not powered for efficacy no statistical analysis was performed
Time Frame: Baseline, Month 6
Population: as for outcome 1
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Particpants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of particpants with Adverse events as a measure of safety and tolerability
Time Frame: 6 months
Population: The safety set consists of all subjects who received at least one dose of study medication. Subjects will be analyzed according to the treatment received.
Measure: Number; unit: Participants
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Number analyzed (Participants) | 6 | 8 | 8 | 6
Participants
  Adverse Events (AE) | 1 | 3 | 3 | 2
  Death | 0 | 0 | 0 | 0
  Non-Fatal Seriuos Aderse Event (SAE) | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Description: The safety set consists of all subjects who received at least one dose of study medication. Subjects were analyzed according to the treatment received.
Arm/Group | AIN457 15 mg/kg | AIN457 7 mg/kg | AIN457 3 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 3/8 | 3/8 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 15 mg/kg (N=6) | AIN457 7 mg/kg (N=8) | AIN457 3 mg/kg (N=8) | Placebo (N=6)
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 15 mg/kg (N=6) | AIN457 7 mg/kg (N=8) | AIN457 3 mg/kg (N=8) | Placebo (N=6)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to early termination this trial was not powered for efficacy no statistical analysis was performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis doesn not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e. data from all sites) in the clinical trial or disclosure of the trial results in their entirety.